CLINICAL TRIAL: NCT05613790
Title: Effect of High-Definition Transcranial Direct Current Stimulation (HD-tDCS) on Attentional Control: an fMRI Study on Healthy Participants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, Afra Souki, Principal Investigator, University of Tehran
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 511098020
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers
Keywords: High-Definition Transcranial Direct Current Stimulation; HD-tDCS; functional Magnetic Resonance Imaging; Attentional control; Attention Network Test

STUDY DESIGN:
Intervention Model Description: Participants are allocated to one of two conditions: Active or Sham.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple-blind study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active HD-tDCS (Experimental): Participants in the active arm will receive 20 min of real High-Definition transcranial direct current stimulation. Additional ramp-up and ramp-down phases at the beginning and the end of stimulation will last for 30 s.
  Interventions: Device: Active High-Definition Transcranial Direct Current Stimulation (HD-tDCS)
- Sham HD-tDCS (Experimental): During the sham session, the montage will be identical, however, the current amplitude will ramp up for 30 seconds, and for the remaining stimulation time, the current flow will terminate and will be kept to zero. Ramp-down phase at the end of stimulation will last for 30 s.
  Interventions: Device: Sham High-Definition Transcranial Direct Current Stimulation (HD-tDCS)

INTERVENTIONS:
Device: Active High-Definition Transcranial Direct Current Stimulation (HD-tDCS) — Portable multi-channel tES stimulation (Starstim 8, Neuroelectric, Barcelona, Spain) will be used.
  Arms: Active HD-tDCS
Device: Sham High-Definition Transcranial Direct Current Stimulation (HD-tDCS) — Portable multi-channel tES stimulation (Starstim 8, Neuroelectric, Barcelona, Spain) will be used.
  Arms: Sham HD-tDCS

SUMMARY:
In a randomized, triple-blind, sham-controlled clinical trial, we will assess the effect of a single session frontal cortex High-Definition transcranial Direct Current Stimulation (HD-tDCS) on brain activity and functional connectivity underlying the behavioral change in attentional control in healthy participants. Participants will be recruited after meeting the inclusion criteria and will be randomly assigned to active or sham stimulation groups. All participants will undergo resting-state functional Magnetic Resonance Imaging (rsfMRI) scan and perform an Attention Network Test (ANT) in a functional Magnetic Resonance Imaging (fMRI) scanner before and after receiving a single session of active or sham HD-tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed healthy adults
* Age range 20-39 years
* Normal or corrected-to-normal vision
* Willing and capable of following study protocol requirements given in the informed consent

Exclusion Criteria:

* Psychiatric conditions (e.g., depression and generalized anxiety disorder, etc.)
* Medical illness or neurological disorder (e.g., cardiovascular illness, anemia, respiratory illness, neurological illness, seizure, etc.)
* Current abuse of drugs or alcohol
* Any conditions that prevent undergoing an fMRI scan or tDCS stimulation according to the fMRI and tDCS safety checklists

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in Attention Network Test (ANT) performance before and after the intervention (active versus sham HD-tDCS) | Immediate before and immediate after intervention
Change in resting state functional connectivity before and after the intervention (active versus sham HD-tDCS) | Immediate before and immediate after intervention
Change in task-based functional connectivity during Attention Network Test (ANT) before and after the intervention (active versus sham HD-tDCS) | Immediate before and immediate after intervention
Change in the blood-oxygen-level-dependent (BOLD) signal during Attention Network Test (ANT) before and after the intervention (active versus sham HD-tDCS) | Immediate before and immediate after intervention

SECONDARY OUTCOMES:
Side effect checklist for transcranial Direct Current Stimulation (Reported as Yes or No) | One day after simulation session

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No